CLINICAL TRIAL: NCT03162926
Title: An Open-Label Study Evaluating the Safety and Tolerability of VC-02™ Combination Product in Subjects With Type 1 Diabetes Mellitus
Brief Title: A Safety and Tolerability Study of VC-02™ Combination Product in Subjects With Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViaCyte (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VC02-102
Record Dates: First submitted 2017-05-19; First posted 2017-05-22 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single-group (Experimental): Up to six (6) VC-02-20 implants
  Interventions: Combination Product: VC-02 Combination Product (aka PEC-Direct)

INTERVENTIONS:
Combination Product: VC-02 Combination Product (aka PEC-Direct) — PEC-01 cells loaded into a Delivery Device

SUMMARY:
The purpose of this trial is to test if VC-02™ combination product can be implanted subcutaneously in subjects with Type 1 Diabetes and maintained safely for up to four (4) months.

ELIGIBILITY:
Inclusion Criteria:

* Men and non-pregnant women of non-childbearing potential
* Diagnosis of T1DM for a minimum of five (5) years
* Stable diabetic treatment
* Willingness to use a continuous glucose meter
* Acceptable candidate for implantation

Exclusion Criteria:

* History of islet cell, kidney, and/or pancreas transplant.
* Two (2) or more severe, unexplained hypoglycemic events within six (6) months of enrollment
* Uncontrolled or untreated thyroid disease or adrenal insufficiency
* Diabetic complications such as severe kidney disease or renal dysfunction, proliferative retinopathy, diabetic foot ulcers, amputations attributable to diabetes, and/or severe peripheral neuropathy
* Non-compliance with current anti-diabetic regimen

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2018-02-15 (Actual)

PRIMARY OUTCOMES:
Incidence of all adverse events reported for subjects | Thru the Month 4 Visit]

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada